CLINICAL TRIAL: NCT02916719
Title: Monitoring of Breast Cancers Treated by Neoadjuvant Radiotherapy Via Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Mieke Cannie, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-PreopBreast-IRM
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: neo-adjuvant radiotherapy; breast cancer; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neo-adjuvant radiotherapy (Experimental): Group of women having undergone a neo-adjuvant radiotherapy for early breast cancer.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI examination after the neo-adjuvant radiotherapy, but before the surgical treatment

SUMMARY:
Magnetic resonance imaging (MRI) is the method of choice in breast cancer to perform the loco-regional staging and direct the treatment.

European Guidelines (EUSOMA) currently recommend MRI for initial evaluation and assessement of the neoadjuvant chemotherapy (NAC) response, for breast cancer. The standard of care consists of realizing a MRI before the start of the NAC and another one after it's ended, six months later.

There is currently no consensus on the realization of an interval MRI for early assessment of the chemosensitivity of the tumor. It would allow though alterations in the therapeutic regimen in the event of a non response. Similarly, there is no consensus on when this interval MRI should be performed.

Some recent studies suggest that Diffusion-weighted Magnetic Resonance Imaging is interesting for the evaluation of the early response. However, these are preliminary studies with quantitative measures realized by the region of interest (ROI) method. A response to neoadjuvant chemotherapy results in elevated values of apparent diffusion coefficients (ADC).

There is'nt any published data on the potential interest of breast MRI after a radiotherapy treatment and before the surgical treatment.

Therefore, the expected benefits of this study are:

* to monitor the early modifications of the perfusion and diffusion parameters at the level of the tumor after radiotherapy, and correlate them to the histology of the surgical monster.
* to assess if MRI is able to objectivate the early signs of response after a radiotherapy neo-adjuvant treatment of breast cancer.

This record is linked to the NCT02858934 record and will share the same cohort of patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological diagnosis of unifocal invasive breast carcinoma, no special type (ductal carcinoma)
* Tumor Staging: cT1-2N0M0
* Luminal A or B
* Candidate for breast conserving surgery
* N0-status confirmed by lymph node cytology

Exclusion Criteria:

* Multifocal/multicentric disease
* Prior thoracic radiotherapy
* Pregnancy
* SBR3 grading
* Triple negative status which benefit neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Anatomo-pathology classification - histological type | Between 2 to 8 days after last radiotherapy session
  The histological type of the tumor will be determined by the Anatomo-Pathology Department of the CHU Brugmann hospital, according to standard of care. The determination will be performed on the initial biopsy samples used for diagnosis and/or on the surgical specimen
Apparent diffusion coefficient (ADC) (mm2/sec) | Baseline (before radiotherapy)
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.
Apparent diffusion coefficient (ADC) (mm2/sec) | Between 2 to 8 days after last radiotherapy session
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No